CLINICAL TRIAL: NCT00903526
Title: Prevalence and Epidemiology of Nosocomial Candidaemia and Antifungal Susceptibility Patterns in an Italian Tertiary-Care Hospital
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Dr Giovanni Guaraldi/ Dr Mauro Codeluppi, Infectoius Disease Clinic
Other Study IDs: 3423/CE
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Candidemia
Keywords: fungal susceptibility
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- candidemia

SUMMARY:
During the past two decades, the frequency of invasive fungal infections has increased dramatically in hospitalised patients throughout the world, and Candida has now emerged as one of the leading causes of bloodstream infections (BSIs). Risk-factors for invasive candidiasis include improvements in intensive care strategies (i.e., central venous catheters, mechanical ventilation, hyper-alimentation), prolonged stays in intensive care units (ICUs), the development of more aggressive surgical techniques, and the prolongation of survival of critically-ill patients. Two other important factors, observed mainly in cancer patients, are colonization of mucous membranes by yeasts, and neutropenia, resulting from increased use of antibiotics and anti-neoplastic agents, respectively. The crude mortality rate of candidaemia is high (38-75%), and the attributable mortality has been estimated at 25-38%. During the past 15 years, the prevalence of infections caused by non-albicans Candida spp. has increased exponentially, so that these organisms now account for > 50% of episodes of fungaemia in various surveys. The increase in invasive fungal infections, the associated high mortality rate, and the emergence of antifungal resistance, have all driven the search for more potent antifungal drugs. The aims of the present study are to investigate the prevalence and the epidemiology of candidaemia and to determine the antifungal susceptibility patterns of Candida spp. isolates from a tertiary-care hospital in Italy.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with a nosocomial candidaemia at the University Hospital of Modena, Italy, between January 1998 and March 2008

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with a nosocomial candidaemia at the University Hospital of Modena, Italy, between January 1998 and March 2008
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-03

PRIMARY OUTCOMES:
The aims of the present study are to investigate the prevalence and the epidemiology of candidaemia and to determine the antifungal susceptibility patterns of Candida spp. isolates from a tertiary-care hospital in Italy. | 2009